CLINICAL TRIAL: NCT04008654
Title: Implementation of ERAS Protocol in Patients Undergoing Surgery for Urinary Incontinence or Pelvic Organ Prolapse
Brief Title: Evaluation of the Benefits of Enhanced Recovery After Surgery (ERAS) Protocol in Pelvic Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Huseyin Kiyak, Principal Investigator, M.D., Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Huseyin2
Record Dates: First submitted 2019-06-30; First posted 2019-07-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Urinary Incontinence; Pelvic Organ Prolapse
MeSH Terms: conditions — Urinary Incontinence; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Active Comparator): This groups will receive ERAS protocol
  Interventions: Behavioral: ERAS Protocol
- Conventional care (Placebo Comparator): This group will not receive the ERAS protocol.
  Interventions: Behavioral: Conventional care

INTERVENTIONS:
Behavioral: ERAS Protocol — Preoperative measures:
  Counseling before hospital admission Fluid, and carbohydrate loading Avoiding prolongation of the fasting period Avoiding bowel preparation or its application only in selective cases Application of antibiotic prophylaxis Application of thromboprophylaxis Avoiding premedication
  Intraoperative measures:
  Use of short-acting anesthetic agents Application of midthoracic, epidural anesthesia/analgesia Refraining from using drains Refraining from salt, and water overload Maintenance of normothermia (heating the body, and use of warmed up intravenous fluids)
  Postoperative:
  Application of midthoracic, epidural anesthesia/analgesia Refraining from use of nasogastric tube Prevention of nausea, and vomiting Refraining from salt, and water overload Earlier removal of catheters Initiation of oral intake at an early period Use of nonopioid oral analgesics/NSAIDs Early mobilization Adherence to the protocol, and auditing results
  Arms: ERAS group
Behavioral: Conventional care — This group of patients will not receive the specific ERAS protocol but will receive conventional care.
  Arms: Conventional care

SUMMARY:
ERAS protocols have been shown to improve recovery in terms of reduced pain, shortened time to ambulation and length of hospital stay. This study aims to investigate the impact of ERAS protocol on time to mobilization and length of hospital stay in patients undergoing surgery for urinary incontinence and pelvic prolapse.

DETAILED DESCRIPTION:
ERAS protocols containing several preoperative, intraoperative and postoperative measures have been shown to improve recovery in terms of reduced pain, shortened time to ambulation and length of hospital stay in patients undergoing surgery. However, data concerning the role of ERAS protocols in urogynecological surgery is limited. The present study, therefore, aimed to address the role of ERAS protocols in patients undergoing surgery for urinary incontinence and pelvic prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled for surgery because of urinary incontinence or pelvic organ prolapse

Exclusion Criteria:

* Insulin dependent diabetes

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Ambulation | Up to 1 week
  Time to ambulation
Hospital stay | Up to 1month
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Kiyak, MD, Principal Investigator — Kanuni Sultan Suleyman Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No